## Official Title:

A Study in Adults on Pre-LT Dialysis With Basiliximab, Delayed Tacrolimus (TAC), Mycophenolate (MMF), and Steroids (Group 1) vs. Basiliximab, Delayed TAC, MMF, Steroids, With Everolimus 30 Days Post-LT (Group 2) vs. TAC, MMF, and Steroids (Group 3)

## **NCT Number:**

NCT04104438

## **Document Date:**

September 3, 2020

## **Statistical Analysis**

Continuous variables were expressed as median (range) and were compared using the Mann-Whitney U test. Categorical variables were expressed as a numerical percentage and compared by the Chi-square test or the Fishers Exact Test. Survival curves were generated by the Kaplan–Meier method, and differences in survival rates were analyzed using the Log-Rank test. All tests were two-sided, and the significance level was p<0.05. All analyses were performed using IBM® SPSS® Statistics version 26 (IBM Corporation, Armonk, NY).